CLINICAL TRIAL: NCT06094790
Title: An Open-Label, Repeat-Dose Study to Evaluate the Pharmacokinetics of Orally Administered CORT125134 Using the Current Capsule Formulation in Healthy Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of the Current Capsule Formulation of CORT125134 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CORT125134-453
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — relacorilant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Subjects will receive CORT125134 150 mg once daily for 14 days
  Interventions: Drug: CORT125134 150 mg
- Cohort 2 (Experimental): Subjects will receive CORT125134 250 mg once daily for 14 days
  Interventions: Drug: CORT125134 250 mg
- Cohort 3 (Experimental): Subjects will receive CORT125134 once daily for 14 days at a dose level decided based on evaluation of steady state exposure from Cohorts 1 and 2
  Interventions: Drug: CORT125134 dose to be determined
- Cohort 4 (optional) (Experimental): Subjects will receive CORT125134 once daily for 14 days at a dose level decided based on evaluation of steady state exposure from Cohorts 1, 2, and 3, if it is considered that this cohort would aid achievement of the study objectives
  Interventions: Drug: CORT125134 dose to be determined

INTERVENTIONS:
Drug: CORT125134 150 mg — CORT125134 150 mg (3 X 50 mg current capsule formulation)
  Arms: Cohort 1
Drug: CORT125134 250 mg — CORT125134 250 mg (5 X 50 mg current capsule formulation)
  Arms: Cohort 2
Drug: CORT125134 dose to be determined — CORT125134 current capsule formulation, dose to be determined
  Arms: Cohort 3; Cohort 4 (optional)

SUMMARY:
A study designed to characterize the plasma pharmacokinetic (PK) profile of CORT125134 in healthy subjects receiving once-daily oral administration of the current capsule formulation of CORT125134 for 14 days.

DETAILED DESCRIPTION:
Initially, subjects will be enrolled into 2 cohorts each of 8 subjects (Cohort 1 and Cohort 2) to receive CORT125134 at 150 mg or 250 mg, respectively. Data from Cohorts 1 and 2 will be evaluated to select dose levels for Cohort 3 and optional Cohort 4.

The secondary objective of the study is to characterize the plasma PK profile of CORT125134 metabolites in healthy subjects receiving once-daily oral administration of the current capsule formulation of CORT125134.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent
* Be healthy males or non-pregnant, non-lactating healthy females
* Must agree to use an adequate method of contraception as described in the study protocol
* Have a body mass index (BMI) of 18 to 32 kg/m^2, inclusive and body weight more than 50 kg (110 pounds)
* Be willing to comply with study restrictions as described in study protocol
* Be able to comply with the requirements of the entire study
* Be judged to be in good health, based on the results of medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory findings
* Have suitable veins for multiple venipuncture/cannulation

Exclusion Criteria:

* Be an employee or immediate family member of the Clinical Research Unit or Corcept
* Have been previously enrolled in this study
* Have multiple drug allergies, or be allergic to any of the components of study drug
* Have a condition that could be aggravated by glucocorticoid blockade (eg, asthma, any chronic inflammatory condition)
* In the 1 year before study drug administration, have a history of drug or alcohol abuse
* In the 6 calendar months before study drug administration, on average: have smoked more than 5 cigarettes/day, consumed more than 14 units (female) or 21 units (male) of alcohol/week (1 unit/drink = 5 ounces of wine, or 12 ounces of beer, or 1.5 ounces of hard liquor), consumed licorice or other glycyrrhetic acid derivatives regularly, in the judgement of the Investigator
* In the 2 calendar months before study drug administration, have donated/ lost blood or plasma in excess of 400 mL
* In the 30 days before study drug administration, have participated in another clinical trial of a new chemical entity or a prescription medicine
* Have a positive test for alcohol or drugs of abuse at Screening or admission
* Have a positive test for exogenous glucocorticoids at Screening
* Have clinically-relevant abnormal findings on vital signs, physical examination, laboratory screening tests, or 12-lead ECG, at Screening and/or before first dose
* Have any medical or social reasons for not participating in the study raised by their primary care physician
* Have any other condition that might increase the risk to the individual or decrease the chance of obtaining satisfactory data, as assessed by the Investigator
* Have taken any prohibited prior medication, as described in study protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-11-15 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve over a dose-interval of plasma CORT125134 (AUCtau) | Predose and at serial timepoints over a dose-interval following dosing on Days 1, 7, and 14
Maximum concentration of plasma CORT125134 (Cmax) | Predose and at serial timepoints up to 24 hours following Day 1 and Day 7 dosing, and at serial timepoints up to 120 hours following Day 14 dosing
AUC from the time of dosing until 24 hours later of plasma CORT125134 (AUC0-24h) | Predose and at serial timepoints up to 24 hours following dosing on Days 1, 7, and 14.
  Statistical analysis of these data will be used to estimate the highest oral dose of CORT125134 current capsule formulation steady state AUC0-24h of plasma CORT125134.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Moraitis, Study Director — Corcept Therapeutics
Locations (1):
- Quotient Sciences, Miami, Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No